CLINICAL TRIAL: NCT06827561
Title: The Effect of Presbyphagia on Urinary Incontinence and Quality of Life in Healthy Elderly People in Nursing Homes
Acronym: Presbyphagia
Status: Completed | Type: Observational
Sponsor: Isparta University of Applied Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: postdr1
Record Dates: First submitted 2025-01-31; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-09

CONDITIONS: Presbyphagia; Incontinence, Urinary; Quality of Life
Keywords: Presbyphagia; Urinary Incontinence; Quality of Life
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Presbyphagia Group: This is a group of elderly people with swallowing disorders. Urinary incontinence and quality of life will be evaluated diagnostically.
- Non-Presbyphagia Group: This group is an elderly group in which swallowing disorder is not detected. Urinary incontinence and quality of life will be evaluated diagnostically.

SUMMARY:
Urinary incontinence in the elderly and health-related quality of life due to urinary incontinence is a common problem in nursing homes. Another problem that occurs in elderly individuals is swallowing disorder. Swallowing disorders that occur with aging are called presbyphagia. Additional health problems such as impaired fluid intake balance, fetal incontinence and sarcopenia may occur after presbyphagia. However, the effect of presbyphagia on urinary incontinence is not known. In this study, we aimed to determine the effect of presbyphagia on urinary incontinence and quality of life in healthy elderly individuals living in a nursing home.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been living in the nursing home for at least 1 year and volunteer to participate in the study
* a mini metal test score of 24 and above

Exclusion Criteria:

* Those who cannot provide information on urinary function and quality of life,
* Those with a history of disease and surgery with mechanisms directly related to swallowing and urinary incontinence,
* Those with a mini mental test score of 23 or less were excluded

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy elderly people living in a nursing home
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Determining the presence of urinary incontinence | 1 day
  Determination of urinary incontinence in the elderly with swallowing problems using the International Consultation on Incontinence Questionnaire Short (ICIQ) scale.
Determining the presence ofquality of life | 1 day
  Determination of health-related quality of life related to urinary incontinence in elderly people with swallowing problems using King's Health Questionnaire (KHQ) scale

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Haci Ahmet Şençopur Huzurevi Yaşli Bakim Ve Rehabilitasyon Merkezi, Uluborlu, Isparta
  - Uluborlu Gardenia Care Center, Uluborlu, Isparta

IPD SHARING:
Plan to Share IPD: No
Sharing the personal data of elderly residents of the institution constitutes a crime for the Republic of Turkey.

REFERENCES:
- [Background] Kakehi S, Wakabayashi H, Isono E, Takemura R, Sato Y, Otsuka Y, Nagai T, Nishioka S, Momosaki R. Association between sarcopenia and urinary dysfunction in patients with dysphagia. Arch Gerontol Geriatr. 2024 Dec;127:105577. doi: 10.1016/j.archger.2024.105577. Epub 2024 Jul 19. PMID 39032316